CLINICAL TRIAL: NCT06440031
Title: Culturally-adapted Manual-assisted Psychological Intervention (CaMaPi) for Adolescents/Young People With a History of Self-harm and Suicidal Ideation in Jos, Nigeria
Brief Title: CaMaPi for Adolescents/Young People With a History of Self-harm and Suicidal Ideation in Jos, Nigeria
Acronym: CaMaPi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: University of Manchester (Other); Jos University Teaching Hospital (Other); Teesside University (Other)
Responsible Party: Principal Investigator, Dr Dung Jidong, PhD, Dr, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0001-5034-0335f
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Self-harm; Suicidal Ideation
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaMaPi (Experimental)
  Interventions: Behavioral: CaMaPi
- TAU (Active Comparator)
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: CaMaPi — CaMaPi is a manually assisted brief psychological intervention that is based on the principles of Cognitive Behaviour Therapy (CBT). The intervention includes psycho-education and a comprehensive cognitive behavioural assessment of the suicidal ideation and self-harm attempt using virtual stories of four young people to be delivered in 8-10 sessions for over three months
  Arms: CaMaPi
Other: TAU — Treatment as Usual (TAU) is routine care, such as diagnosis, assessment, psychotherapy, monitoring and any form of intervention (e.g., medication prescription) available at the collaborating service.
  Arms: TAU

SUMMARY:
Suicide and self-harm are global disease burden that contributes significantly to years of lost life and mortality.

DETAILED DESCRIPTION:
Self-harm and suicidal ideation represent a significant global public health concern (Knipe et al., 2022), affecting about 14.6 million people yearly (Nichols et al., 2021). Globally, over 700 000 people die by suicide annually (World Health Organization -- WHO, 2023).

Suicide is the fourth leading cause of death among 15-29-year-olds, and 77% of global suicides occur in low- and middle-income countries, including Nigeria (WHO, 2023). The psychological impact of suicidal ideation includes continuing high tendencies of self-harm (Jidong et al., 2024).

Despite the increasing rates of suicide and self-harm in Nigeria, this topic is understudied, with no culturally appropriate or sustainable psychological interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16-24 years presenting to the participating services, and emergency departments or admitted after an episode of self-harm to the participating hospitals or self-referrals.
* Participants will have to be living within the catchment area of the participating practices, services and hospitals.
* Not needing inpatient psychiatric treatment.

Exclusion Criteria:

* Severe mental illness (such as Psychotic disorder).
* Conditions limiting engagement with assessment/intervention.
* Temporary resident unlikely to be available for follow up.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in acceptance and satisfaction with the intervention | Change is being assessed from baseline, end of intervention at 12 weeks, and at 12 weeks post-intervention
  Primary outcome measure would be assessed using the Service Satisfaction Scale

SECONDARY OUTCOMES:
Change in suicidal ideation | Change is being assessed from baseline, end of intervention at 12 weeks, and at 12 weeks post-intervention
  Secondary outcome measure would be assessed using the Beck Scale for Suicide Ideation
Change in hopelessness | Change is being assessed from baseline, end of intervention at 12 weeks, and at 12 weeks post-intervention
  Secondary outcome measure would be assessed using the Beck Hopelessness Scale
Change in Health Status | Change is being assessed from baseline, end of intervention at 12 weeks, and at 12 weeks post-intervention
  Secondary outcome measure would be assessed using the EQ-5D-5L quality of health scale
Change in repetition rate's of self-harm | Change is being assessed from baseline, end of intervention at 12 weeks, and at 12 weeks post-intervention
  Secondary outcome measure would be assessed using an adapted Suicide Attempt Self-Injury Interview
Change in use of health services | Change is being assessed from baseline, end of intervention at 12 weeks, and at 12 weeks post-intervention
  Secondary outcome measure would be assessed using Client Service Receipt Inventory
Change in psychological distress | Change is being assessed from baseline, end of intervention at 12 weeks, and at 12 weeks post-intervention
  Secondary outcome measure would be assessed using Kessler Psychological Distress Scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jidong DE, Ike TJ, Taru MY, Pwajok JY, Nwoga CN, Jidong JE, Mwankon SB, Francis C, Husain N. Culturally Adapted Manual-Assisted Psychological Intervention (CaMaPI) for Adolescents/Young People With a History of Self-Harm and Suicidal Ideation in Nigeria: A Randomised Controlled Feasibility Trial. Clin Psychol Psychother. 2025 May-Jun;32(3):e70098. doi: 10.1002/cpp.70098. PMID 40497640